CLINICAL TRIAL: NCT01339598
Title: Remediation of Cognitive Dysfunction in Euthymic Bipolar Disorder Patients Using Transcranial Direct Current Stimulation (tDCS)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of New South Wales (Other)
Responsible Party: Dr Donel Martin, University of New South Wales
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: HREC 11065
Record Dates: First submitted 2011-04-07; First posted 2011-04-20 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-07

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sham transcranial direct current stimulation (Sham Comparator)
  Interventions: Device: Transcranial direct current stimulation (Eldith DC Stimulator)
- Transcranial direct current stimulation (Active Comparator)
  Interventions: Device: Transcranial direct current stimulation (Eldith DC Stimulator)
- Different transcranial direct current stimulation montage (Active Comparator)
  Interventions: Device: Transcranial direct current stimulation (Eldith DC Stimulator)

INTERVENTIONS:
Device: Transcranial direct current stimulation (Eldith DC Stimulator) — Eldith DC Stimulator (NeuroConn GmbH, Germany)

SUMMARY:
This study aims to investigate the potential for Transcranial Direct Current Stimulation (tDCS) to enhance cognitive functioning in euthymic bipolar patients through comparing the effect of active or sham tDCS (placebo control) during the performance of two cognitive tasks. The investigators hypothesize that task performance will be improved with active relative to sham tDCS.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be right-handed subjects aged 18-65 meeting DSM-IV diagnostic criteria for bipolar disorder, with no acute episodes of depression or mania within the previous 12 weeks
* A score of ≤ 20 on the MADRS, and a score of ≤ 6 on the YMRS, who have been on a stable dose of mood stabiliser medications for at least 1 month.

Exclusion Criteria:

* Patients with high suicide risk
* Co-morbid DSM-IV diagnosis of any psychotic disorder (current or within the last year), schizophrenia and schizoaffective disorder
* Mental retardation
* A history of drug or alcohol abuse or dependence within the last 3 months
* Co-morbid attention deficit hyperactivity disorder (ADHD), or any neurological disorder
* Recent stroke
* Head injury
* History of seizure, or who have had electroconvulsive therapy (ECT) within the 6 months preceding enrolment.
* Participants will also be excluded if currently taking medications known to be associated with frank cognitive impairment (e.g., benzodiazepines).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-09; Primary Completion 2014-12 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Total correct responses. | Across each session (approximately 1 hour in duration), with each session conducted at least 1 week apart.
  Total number of correct responses on each task in each session.

CONTACTS AND LOCATIONS:
Locations (1):
- University of New South Wales, Sydney, New South Wales, Australia